CLINICAL TRIAL: NCT04778072
Title: A Randomised, Double-blinded, Parallel Group Study to Demonstrate the Adherence and Efficacy of Different Doses of Iron Supplement in Subjects With or At-risk of Iron Deficiency With a History of Intolerance to Oral Iron
Brief Title: A Clinical Study on Adherence and Efficacy of Different Doses of Active Iron in Treatment Resistant Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Solvotrin Innovations Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFCRO-80
Record Dates: First submitted 2021-02-26; First posted 2021-03-02 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Premenopause; Iron-deficiency; Iron Adverse Reaction; Iron Deficiency Anemia; Heavy Menstrual Bleeding
Keywords: Randomised controlled trial; Double blind; Ferrous sulfate; Intolerance; Oral iron; Adherence; Efficacy; Whey protein; Active Iron
MeSH Terms: conditions — Anemia, Iron-Deficiency; Menorrhagia | interventions — ferrous sulfate

STUDY DESIGN:
Intervention Model Description: Three groups in parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomized into one of three arms (20 subjects per arm) but will be blinded as to which group they are in. The three arms are as follows:
  Group 1: ACTIVE IRON™ (ferrous sulfate) 14 mg elemental iron once daily (and matching placebo) Group 2: ACTIVE IRON™ (ferrous sulfate) 25 mg elemental iron once daily (and matching placebo) Group 3: ACTIVE IRON™ (ferrous sulfate) 25 mg elemental iron twice daily (and matching placebo)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): ACTIVE IRON™ (ferrous sulfate) 14 mg elemental iron once daily with matching placebo
  Interventions: Dietary Supplement: Ferrous sulfate 14mg once daily
- Group 2 (Experimental): ACTIVE IRON™ (ferrous sulfate) 25 mg elemental iron once daily with matching placebo
  Interventions: Dietary Supplement: Ferrous sulfate 25mg once daily
- Group 3 (Experimental): ACTIVE IRON™ (ferrous sulfate) 25 mg elemental iron twice daily with matching placebo
  Interventions: Dietary Supplement: Ferrous sulfate 25mg twice daily

INTERVENTIONS:
Dietary Supplement: Ferrous sulfate 14mg once daily — ACTIVE IRON™ (ferrous sulfate) 14 mg elemental iron once daily with matching placebo
  Other Names: ACTIVE IRON™
  Arms: Group 1
Dietary Supplement: Ferrous sulfate 25mg once daily — ACTIVE IRON™ (ferrous sulfate) 25 mg elemental iron once daily with matching placebo
  Other Names: ACTIVE IRON™
  Arms: Group 2
Dietary Supplement: Ferrous sulfate 25mg twice daily — ACTIVE IRON™ (ferrous sulfate) 25 mg elemental iron twice daily
  Other Names: ACTIVE IRON™
  Arms: Group 3

SUMMARY:
A randomized, placebo controlled, parallel group, double blind study to compare the 3-month adherence and efficacy of Active Iron in subjects with or at-risk of iron deficiency and a history of intolerance to oral iron. Subjects with intolerance and treatment failure due to oral iron (male and female subjects, aged 18 to 55 years, with mild to moderate iron deficiency, with or without anaemia) are eligible. Sixty subjects are randomised into three groups (14 mg elemental iron, 25mg elemental iron and 50mg elemental iron daily). The primary objective is to assess adherence/persistence (including using pill counts). Secondary objectives are to assess gastrointestinal tolerability, haematological efficacy and health related quality of life.

DETAILED DESCRIPTION:
More than 2.2. billion people worldwide have anaemia and half of this burden is caused by iron deficiency [Lopez 2016]. The commonest causes of iron deficiency are inadequate intake, poor absorption of iron [Stoffel 2017] and blood loss, for example due to menstruation [World Health Organization Guideline: Daily iron supplementation in adult women and adolescent girls; Geneva 2016, Low 2016]. Supplementation with oral iron is well established to prevent and treat iron deficiency anaemia and to promote recovery of iron and haemoglobin levels post blood loss or blood donation [Low 2016, McNamee 2013]. However, iron food fortification and oral iron supplements are frequently limited by poor absorption and poor tolerability [Munoz 2009]. Ferrous sulfate is considered the gold standard and the only oral iron form on the WHO Essential Medicines List, yet has fractional absorption of only 16%-21% from daily or alternative daily doses [Stoffel et al 2017]. It is also poorly tolerated, causing adverse GI effects in a majority of patients [Pereira 2014]. This results in poor adherence in up to 50% of users, significant nutritional deficit and treatment failure [Tolkien 2015]

We have previously evaluated a formulation of microspheres of iron sulfate in a denatured whey protein (WP) matrix at a daily elemental iron dose of 25mg daily, marketed as Active Iron, in comparison with equi-dose immediate release and modified release ferrous sulfate (Wang et al. Acta Haematologica Acta Haematol 2017;138:223-232). In these evaluations, the iron-WP formulation has shown better absorption and there were no reports of adverse effects. Furthermore, in-vitro data show that the iron-WP matrix formulation can protect HT20 gut endothelial cells and CaCO2 cells from oxidative stress and cell damage associated with ferrous sulfate. In a post-marketing survey of 101 people taking Active Iron (age 43 ± 10 years, 83% female) with a history of intolerance to oral iron, 87% reported no adverse effects after 2 weeks.

Therefore, the present study aims to compare the 3-month adherence and efficacy associated with a 25mg single daily dose, a lower (14mg) single daily dose and twice daily dosing with 25mg (50mg daily), in subjects with treatment failure (iron deficiency and with a history of intolerance to oral iron). The primary objective of the study is to assess the proportion of subjects adherent and persistent (>80% based on pill counts) from baseline to weeks 6 and baseline to week 12. Secondary objectives aim to further assess compliance (average compliance), tolerability (incidence of gastrointestinal symptoms GSRS instrument), efficacy (change in haemoglobin, ferritin, transferrin saturation, iron binding protein) and health related quality of life (SF36 instrument).

At least 90 subjects will be screened in order to identify up to 60 eligible subjects, and 54 evaluable subjects. Participants will be male and female, between 18 and 55 years of age, with mild to moderate iron deficiency anaemia (haemoglobin ≥9.5 g/dL and <12.0 g/dL for females and ≥10.0 g/dL and <13.0 g/dL for males and ferritin < 30 µg/L) or ferritin < 30 µg/L and no anaemia. There will be stratified randomisation to include up to 30 patients with iron deficiency and mild to moderate anaemia as well as up to 30 patients with iron deficiency without anaemia. Other pre-specified sub-groups for evaluation of the primary and secondary endpoints include women with reported symptoms of heavy menstrual bleeding and participants with intolerance of liquid iron products or lower doses (< 50mg elemental iron). Separate analysis of primary and secondary endpoints will be carried out in participants in the multivitamin and mineral sub study. Finally, due to the suspension of some clinics during Covid lockdown, we carried out a prespecified analysis of patients completing the study before the onset of the Covid 19 Pandemic.

Subjects will be randomised to one of three treatment arms:

1. ACTIVE IRON™ (ferrous sulfate) 14 mg elemental iron once daily (plus matching placebo)
2. ACTIVE IRON™ (ferrous sulfate) 25 mg elemental iron once daily (plus matching placebo)
3. ACTIVE IRON™ (ferrous sulfate) 25 mg elemental iron twice daily (plus matching placebo)

The study will involve 4 visits over a 12 to 14-week period. At the screening visit (visit 1), informed consent shall be obtained. Demographic data, vitals, anthropometric measurements and prior and concomitant medications will be recorded. Subjects will be asked questions relating to their iron deficiency anaemia and medical history associated with this. Female subjects will be asked questions regarding their menstrual periods and intolerance to other iron products. A fasting blood sample will be collected and a full blood count, including Ferritin and Serum iron/Transferrin will be measured. Blood and serum samples will be frozen and retained for post-hoc analysis of other biomarkers relevant to iron metabolism (e.g. hepcidin, soluble transferrin receptor).

Once eligibility is confirmed the subject will be invited to attend a baseline visit (visit 2, Time 0). At this visit, a blood sample will be collected and a full blood count, including Ferritin and Serum iron/Transferrin will be measured. For women of childbearing age, a urine sample will be collected, and pregnancy test performed. Subjects will be queried about any changes in their health status and any non-treatment emergent events and medications will be recorded. Subjects will complete the following questionnaires: Gastrointestinal Symptom Rating Scale (GSRS Instrument), the Short Form-36 (SF-36 Instrument) and for women who are menstruating, they will report the date, duration and blood flow of their last menstrual period.

Subjects will be randomized into one of three treatment groups, but will be blinded as to which group they are in. Subjects will be supplied with a 6-week supply of study product and instructions on dosing. Subjects will be instructed to following their habitual diet and exercise routine and to not consume any disallowed medications or supplements that could interfere with the assessment of the study product for the duration of the study. Subjects will be provided with an appointment to return to the study site at week 6.

At week 3 and 9 ('phone visits'), all subjects will be asked (to complete the GSRS, and women who are menstruating, will complete Menstrual Period Questionnaire, to record the date, duration and blood flow of their last menstrual period.

Subjects will return to the clinic site at week 6 (visit 3) and 12 (visit 4). At each visit, subjects will be queried about any changes in their health status and any adverse events and medications will be recorded. A blood sample will be collected and a full blood count, including Ferritin and Serum iron/Transferrin will be measured. Subjects will complete the following questionnaires: GSRS, SF-36 and for women who are menstruating, the Menstrual Period Questionnaire. Subjects will return any unused study product and additional product will be dispensed. The adherence based on pill count will be determined for the period. Subjects will be instructed to continue following their habitual diet and exercise routine and to not consume any disallowed medications or supplements that could interfere with the assessment of the study product for the duration of the study.

At the 4th visit (week 12), subjects will be invited to partake in an optional, open-label, follow-up for 3 months after the completion of the blinded intervention phase. Participants who decide to partake in the optional, open-label follow-up study will continue to receive the same dose of Active Iron™ as they received during the blinded intervention phase, for a further 12 weeks, in addition to a multivitamin and mineral complex that is designed to maximise iron metabolism and haemoglobin/red blood cell formation. This complex contains vitamin A, D, B2, B6, B12, folic acid and copper. Subjects will return for an interim follow-up visit at week 18 (visit 5), and a final visit at week 24 (visit 6). At these visits subjects will undergo standard assessments and complete the following questionnaires: GSRS, SF-36 and for women who are menstruating, the Menstrual Period Questionnaire. Subjects will also answer questions on the tolerability of the study product.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent
2. Be between 18 and 55 years of age
3. Have ferritin levels <30 µg/L
4. Have a history of intolerance to oral iron
5. Have mild to moderate anaemia (haemoglobin ≥9.5 g/dL and <12.0 g/dL for females and ≥10.0 g/dL and <13.0 g/dL for males, up to 30 patients) or no anaemia (up to 30 patients)
6. Be in generally good health as determined by the investigator

Exclusion Criteria:

1. A history of dairy allergy or are hypersensitive to any of the components of the test product,
2. Are currently taking any iron supplements, or have done so in the previous 2 weeks,
3. Current inflammatory bowel disease (Crohn's disease or ulcerative colitis),
4. Severe anemia (females with hemoglobin <9.5 g/dL and males with hemoglobin <10.0 g/dL)
5. Females that have started menopause,
6. Females using extended-cycle birth control pills
7. Have a significant acute or chronic, unstable and untreated disease or any condition, which contraindicates, in the investigator's judgement, entry to the study,
8. Having a condition or have taken a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results; for example, no concurrent medication which interferes with the absorption of iron (e.g. tetracyclines, calcium supplements),
9. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial,
10. Subjects may not be receiving treatment involving experimental drugs. If the subject has been in a recent experimental trial, these must have been completed not less than 30 days prior to this study,
11. Have a malignant disease or any concomitant end-stage organ disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-08 (Actual); Primary Completion 2021-04-09 (Estimated); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects adherent/persistent (6 weeks) | 6 weeks
  To assess the change in proportion of subjects adherent/persistent (>80% based on pill counts) from baseline to week 6
Proportion of subjects adherent/persistant (12 weeks) | 12 weeks
  To assess the change in proportion of subjects adherent/persistant (>80% based on pill counts) from baseline to week 12

SECONDARY OUTCOMES:
Upper gastrointestinal symptoms (12 weeks) | 12 weeks
  To assess the difference in incidence of upper GI symptoms from baseline to 12 weeks
Lower gastrointestinal symptoms (12 weeks) | 12 weeks
  To assess the difference in incidence of lower GI symptoms from baseline to 12 weeks
Change in GSRS (12 weeks) | 12 weeks
  To assess the change in gastrointestinal tolerability using GSRS from baseline to 12 weeks
Change in haemaglobin (12 weeks) | 12 weeks
  To assess the change in haemoglobin from baseline to 12 weeks in those with anaemia
Change in ferritin (12 weeks) | 12 weeks
  To assess the change in ferritin from baseline to 12 weeks
Change in transferrin saturation (12 weeks) | 12 weeks
  To assess the change in transferrin saturation from baseline to 12 weeks
Change in health related quality of life (12 weeks) | 12 weeks
  To assess the change in tiredness and energy HRQOL using SF36 from baseline to 12 weeks

OTHER OUTCOMES:
Median adherence (6 weeks) | 6 weeks
  To assess the median adherence based on pill count from baseline to 6 weeks
Median adherence (12 weeks) | 12 weeks
  To assess the median adherence based on pill count from baseline to 12 weeks
Change in GSRS (6 weeks) | 6 weeks
  To assess the change in gastrointestinal tolerability using GSRS from baseline to 6 weeks
Upper and lower gastrointestinal symptoms (6 weeks) | 6 weeks
  To assess the incidence of upper and lower GI symptoms from baseline to 6 weeks
Change in haemaglobin (6 weeks) | 6 weeks
  To assess the change in hemoglobin from baseline to 6 weeks in those with anaemia
Increase in haemaglobin (to at least 12g/dL in women and 13g/dL in men) (6 weeks) | 6 weeks
  To assess the proportion of subjects with haemoglobin increase to at least 12 g/dL (women) and 13 g/dL (men) from baseline to 6 weeks
Increase in haemaglobin (>1g/dL) (6 weeks) | 6 weeks
  To assess the proportion of subjects with hemoglobin increase >1 g/dL from baseline to 6 weeks
Increase in haemaglobin (to at least 12g/dL in women and 13g/dL in men) (12 weeks) | 12 weeks
  To assess the proportion of subjects with hemoglobin increase to at least 12 g/dL (women) and 13 g/dL (men) from baseline to 12 weeks
Increase in haemaglobin (>1g/dL) (12 weeks) | 12 weeks
  To assess the proportion of subjects with hemoglobin increase >1 g/dL from baseline to 12 weeks
Change in ferritin (6 weeks) | 6 weeks
  To assess the change in ferritin from baseline to 6 weeks
Increase in ferritin (to >12 µg/L) (6 weeks) | 6 weeks
  To assess the proportion of subjects with ferritin > 12 µg/L from baseline to 6 weeks
Increase in ferritin (to >12 µg/L) (12 weeks) | 12 weeks
  To assess the proportion of subjects with ferritin > 12 µg/L from baseline to 12 weeks
Increase in ferritin (to >30 µg/L) (6 weeks) | 6 weeks
  To assess the proportion of subjects with ferritin > 30 µg/L from baseline to 6 weeks
Increase in ferritin (to >30 µg/L) (12 weeks) | 12 weeks
  To assess the proportion of subjects with ferritin > 30 µg/L from baseline to 12 weeks
Change in transferrin saturation (6 weeks) | 6 weeks
  To assess the change in transferrin saturation from baseline to 6 weeks
Change in transferrin saturation (>20%) (6 weeks) | 6 weeks
  To assess the proportion of subjects with transferrin saturation > 20% from baseline to 6 weeks
Change in transferrin saturation (>20%) (12 weeks) | 12 weeks
  To assess the proportion of subjects with transferrin saturation > 20% from baseline to 12 weeks
Change in iron binding protein (6 weeks) | 6 weeks
  To assess the change in iron binding protein from baseline to 6 weeks
Change in iron binding protein (12 weeks) | 12 weeks
  To assess the change in iron binding protein from baseline to 12 weeks
Change in health related quality of life (6 weeks) | 6 weeks
  To assess the change in HRQOL using SF36 from baseline to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shauni Fitzgerald, MSC, Study Director — Atlantia Clinical Trials
Locations (1):
- Atlantia Clinical Trials, Cork, Co Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopez A, Cacoub P, Macdougall IC, Peyrin-Biroulet L. Iron deficiency anaemia. Lancet. 2016 Feb 27;387(10021):907-16. doi: 10.1016/S0140-6736(15)60865-0. Epub 2015 Aug 24. PMID 26314490
- [Background] Low MS, Speedy J, Styles CE, De-Regil LM, Pasricha SR. Daily iron supplementation for improving anaemia, iron status and health in menstruating women. Cochrane Database Syst Rev. 2016 Apr 18;4(4):CD009747. doi: 10.1002/14651858.CD009747.pub2. PMID 27087396
- [Background] McNamee T, Hyland T, Harrington J, Cadogan S, Honari B, Perera K, Fitzgerald AP, Perry IJ, Cahill MR. Haematinic deficiency and macrocytosis in middle-aged and older adults. PLoS One. 2013 Nov 7;8(11):e77743. doi: 10.1371/journal.pone.0077743. eCollection 2013. PMID 24244281
- [Background] Munoz M, Villar I, Garcia-Erce JA. An update on iron physiology. World J Gastroenterol. 2009 Oct 7;15(37):4617-26. doi: 10.3748/wjg.15.4617. PMID 19787824
- [Background] Pereira DI, Couto Irving SS, Lomer MC, Powell JJ. A rapid, simple questionnaire to assess gastrointestinal symptoms after oral ferrous sulphate supplementation. BMC Gastroenterol. 2014 Jun 4;14:103. doi: 10.1186/1471-230X-14-103. PMID 24899360
- [Background] Stoffel NU, Cercamondi CI, Brittenham G, Zeder C, Geurts-Moespot AJ, Swinkels DW, Moretti D, Zimmermann MB. Iron absorption from oral iron supplements given on consecutive versus alternate days and as single morning doses versus twice-daily split dosing in iron-depleted women: two open-label, randomised controlled trials. Lancet Haematol. 2017 Nov;4(11):e524-e533. doi: 10.1016/S2352-3026(17)30182-5. Epub 2017 Oct 9. PMID 29032957
- [Background] Tolkien Z, Stecher L, Mander AP, Pereira DI, Powell JJ. Ferrous sulfate supplementation causes significant gastrointestinal side-effects in adults: a systematic review and meta-analysis. PLoS One. 2015 Feb 20;10(2):e0117383. doi: 10.1371/journal.pone.0117383. eCollection 2015. PMID 25700159
- [Derived] Ledwidge M, Ryan F, Seoighe A, Santos-Martinez MJ, Ryan C, Gilmer JGF. Management of iron deficiency in women of childbearing age with oral iron intolerance: a prospective, randomised, controlled trial of three doses of an iron-whey-protein formulation : Prospective RandomisEd study of women of Childbearing age with gastroInteStinal Intolerance to Oral iroN (PRECISION). Int J Clin Pharm. 2024 Apr;46(2):390-400. doi: 10.1007/s11096-023-01640-7. Epub 2023 Dec 26. PMID 38147281